CLINICAL TRIAL: NCT04310514
Title: Effects of Rehydration During Physical Exercise on Acute Kidney Injury Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Wojciech Wolyniec, Principal Investigator, Medical University of Gdansk
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 04-0532/09/776
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Acute Kidney Injury
Keywords: biomarker; albuminuria; uric acid
MeSH Terms: conditions — Acute Kidney Injury; Albuminuria | interventions — Fructose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: glucose - fructose - xylitol - saccharose (Active Comparator): * glucose 35 g (500ml of 7% solution);
  * fructose 35 g (500ml of 7% solution);
  * xylitol 35 g (500ml of 7% solution);
  * saccharose 35 g (500ml of 7% solution)
  Interventions: Dietary Supplement: Fructose/glucose/xylitol/saccharose
- Experimental: fructose - glucose - saccharose - xylitol (Active Comparator): * glucose 35 g (500ml of 7% solution);
  * fructose 35 g (500ml of 7% solution);
  * xylitol 35 g (500ml of 7% solution);
  * saccharose 35 g (500ml of 7% solution)
  Interventions: Dietary Supplement: Fructose/glucose/xylitol/saccharose
- Experimental: xylitol - saccharose - glucose - fructose (Active Comparator): * glucose 35 g (500ml of 7% solution);
  * fructose 35 g (500ml of 7% solution);
  * xylitol 35 g (500ml of 7% solution);
  * saccharose 35 g (500ml of 7% solution)
  Interventions: Dietary Supplement: Fructose/glucose/xylitol/saccharose
- Experimental: saccharose - xylitol - fructose - glucose (Active Comparator): * glucose 35 g (500ml of 7% solution);
  * fructose 35 g (500ml of 7% solution);
  * xylitol 35 g (500ml of 7% solution);
  * saccharose 35 g (500ml of 7% solution)
  Interventions: Dietary Supplement: Fructose/glucose/xylitol/saccharose

INTERVENTIONS:
Dietary Supplement: Fructose/glucose/xylitol/saccharose — 1. Intervention: rehydration with glucose solution. Glucose will be administered at a dose of 35 mg (500 ml of 7% solution) taken orally once, in the middle of soccer training session, at approximately 10.00 a.m.
  2. Intervention: rehydration with fructose solution. Fructose will be administered at a dose of 35 mg (500 ml of 7% solution) taken orally once, in the middle of soccer training session, at approximately 10.00 a.m.
  3. Intervention: rehydration with xylitol solution. Xylitol will be administered at a dose of 35 mg (500 ml of 7% solution) taken orally once, in the middle of soccer training session, at approximately 10.00 a.m.
  4. Intervention: rehydration with sucrose solution Saccharose will be administered at a dose of 35 mg (500 ml of 7% solution) taken orally once, in the middle of soccer training session, at approximately 10.00 a.m.

SUMMARY:
Rehydration during and after physical exercise is essential to avoid acute kidney injury.

Soft drinks are commonly used during exercise. High intake of carbohydrates is leading to obesity and metabolic disorders. Fructose intake is leading to uric acid abnormalities and kidney injury.

30 healthy soccer players will be studied. During four training sessions subjects will intake 500 ml 7% soft drinks containing glucose, fructose, saccharose or xylitol.

Changes in acute kidney injury markers, markers of kidney tubular function as well as changes in CRP, glucose, cholesterol and uric acid levels will be studied..

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* well-trained soccer players
* informed consent

Exclusion Criteria:

* chronic diseases, especially kidney problems
* sigificant changes in urinalysis
* creatinine level above normal values

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in urinary AKI biomarkers (urianry NGAL, urinary KIM -1, urinary cystatin-C) after physical exercise | after 60-90 min of pysical exercise
Changes in fractional uric acid excretion | after 60-90 min of pysical exercise

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Renke, prof, Study Chair — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wolyniec W, Szwarc A, Kasprowicz K, Zorena K, Jaskulak M, Renke M, Naczyk M, Ratkowski W. Impact of hydration with beverages containing free sugars or xylitol on metabolic and acute kidney injury markers after physical exercise. Front Physiol. 2022 Oct 20;13:841056. doi: 10.3389/fphys.2022.841056. eCollection 2022. PMID 36338481